CLINICAL TRIAL: NCT02103335
Title: A Phase 1, Multicenter, Open-label, Dose-Escalation Combination Study of Pomalidomide, Marizomib, and Low-Dose Dexamethasone in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Combination Study of Pomalidomide, Marizomib, and Low-Dose Dexamethasone in Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPI-0052-107
Record Dates: First submitted 2014-03-27; First posted 2014-04-03 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma in Relapse; Refractory Multiple Myeloma; Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; Pomalidomide; Marizomib; Low dose Dexamethasone; Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — pomalidomide; marizomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group Assignment (Experimental): Combination Pomalidomide, low-dose Dexamethasone, and Marizomib:
  Interventions: Drug: pomalidomide; Drug: marizomib; Drug: low-dose dexamethasone

INTERVENTIONS:
Drug: pomalidomide — Oral Pomalidomide, days 1-21 of 28 day cycle, dose 3 to 4 mg
  Other Names: POMALYST
Drug: marizomib — IV Marizomib, 0.2 to 0.5 mg/m2 on days 1, 4, 8, 11 of 28 day cycle
  Other Names: NPI-0052
Drug: low-dose dexamethasone — Oral Dexamethasone, days 1, 2, 4, 5, 8, 9, 11, 12, 15, 16, 22, 23 of 28 day cycle, 5 or 10 mg

SUMMARY:
This is a Phase 1 clinical trial to evaluate a new combination of drugs for the treatment of relapsed or refractory (drug-resistant) multiple myeloma. The drugs being studied are:

* Pomalidomide (POMALYST®) is a drug that affects the immune system (an immunomodulatory drug) that has been approved by the United States (US) Food and Drug Administration (FDA) for the treatment of multiple myeloma.
* Marizomib is an investigational drug being developed by Triphase that is being studied for the treatment of multiple myeloma. Investigational drugs are drugs that have not yet been approved by health authorities, such as the FDA, for general use but have been approved for use in specific clinical studies. Marizomib inhibits a cellular machine called the proteasome, which destroys unnecessary or damaged proteins. Other proteasome inhibitors have been shown to be effective in the treatment of multiple myeloma.
* Dexamethasone is a corticosteroid drug that affects the immune system (an immunomodulatory drug) that has been approved by the FDA for the treatment of multiple myeloma.

This is the first study to evaluate the three-drug combination of pomalidomide (POM), marizomib (MRZ), and dexamethasone (LD-DEX) in humans. Pomalidomide, alone or in combination with dexamethasone, is approved by the FDA for the treatment of relapsed or refractory multiple myeloma.

The primary objective of this study is to determine the best drug dosing levels for this three-drug combination, including the highest safe doses and/or the recommended doses for future clinical studies of this drug combination. The secondary purposes of this study are to determine the safety of this drug combination and its effectiveness in treating relapsed or refractory multiple myeloma. The study will include examination of levels of all three drugs in the blood during various time points during treatment.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following criteria to be eligible for study participation:

1. At least 18 years at the time of signing the informed consent form.
2. Able to understand and voluntarily sign an informed consent form prior to any study-related assessments/procedures.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Documented diagnosis of multiple myeloma and measurable disease by serum or urine protein electrophoresis (SPEP or UPEP): SPEP ≥0.5 g/dL, UPEP ≥200 mg/24 hours, or involved serum free light chain (FLC) level ≥10 mg/dL provided the serum FLC ratio is abnormal.
5. Previously received 1 or more lines of anti-myeloma therapy that must have included both lenalidomide and bortezomib (either separately or in combination).
6. Documented disease progression during or within 60 days after their most recent line of anti myeloma therapy.
7. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.
8. All study participants in the USA must be registered into the mandatory POMALYST REMS™ (Risk Evaluation & Mitigation Strategy) program, and be willing and able to comply with the requirements of the POMALYST REMS™ program.
9. All study participants in the USA who are females of child-bearing potential (FCBP) must adhere to the scheduled pregnancy testing as required in the POMALYST REMS™ program.
10. All study participants outside the USA must agree to comply with the POMALYST® PPRMP requirements.
11. All subjects must be able and agree to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
12. For females of child bearing potential (FCBP): Agree to use 2 reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study treatment, while participating in the study (including dose interruptions), and for at least 28 days after study treatment discontinuation; must follow pregnancy testing requirements as outlined in the POMALYST REMS™ program or the PPRMP.
13. For all females: Agree to abstain from breastfeeding during study participation and for at least 28 days after study treatment discontinuation.
14. For all males: Agree to use a latex or synthetic condom during any sexual contact with FCBP while participating in the study and for at least 28 days following discontinuation from study treatment, even if he has undergone a successful vasectomy.
15. For all males: Agree to refrain from donating semen or sperm while on study and for at least 28 days after discontinuation from study treatment.
16. Refrain from donating blood while on study treatment and for at least 28 days after discontinuation from study treatment.
17. Agree not to share medication.

Exclusion Criteria

Subjects with any of the following will be excluded from participation in the study:

1. Peripheral neuropathy Grade ≥2.
2. Non-secretory multiple myeloma.
3. Any of the following laboratory abnormalities:

   * ANC <1,000/µL;
   * Platelet count <50,000/µL for subjects in whom <50% of bone marrow nucleated cells are plasma cells; or a platelet count <30,000/µL for subjects in whom ≥50% of bone marrow nucleated cells are plasma cells;
   * Creatinine clearance (CrCL) <45 mL/min as measured directly or as calculated according to Cockcroft Gault formula;
   * Corrected serum calcium >13.5 mg/dL (>3.4 mmol/L);
   * Hemoglobin <8 g/dL (<4.9 mmol/L; prior red blood cell [RBC] transfusion or recombinant human erythropoietin use is permitted before study entry);
   * Serum aspartate aminotransferase (AST) >3.0 x upper limit of normal (ULN);
   * Serum alanine aminotransferase (ALT) >3.0 x ULN;
   * Serum total bilirubin >1.5 x ULN (>3.0 x ULN for subjects with known Gilbert's disease).
4. Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥5 years. Subjects may be entered earlier than 5 years if they have received curative treatment for the following:

   * Basal cell carcinoma of the skin;
   * Squamous cell carcinoma of the skin;
   * Carcinoma in situ of the cervix;
   * Carcinoma in situ of the breast;

   Or if they have:

   o Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or non metastatic prostate cancer that is in complete remission or does not require treatment.
5. Previous therapy with POM and/or MRZ.
6. History of allergic reaction or hypersensitivity to thalidomide, lenalidomide, bortezomib, carfilzomib, boron, mannitol, or DEX.
7. Grade ≥3 rash during prior thalidomide or lenalidomide therapy.
8. Gastrointestinal disease that may significantly alter the absorption of POM.
9. History of the following:

   * Congestive heart failure of Class III or IV of the New York Heart Association (NYHA) classification;
   * Myocardial infarction within 12 months prior to starting study treatment;
   * Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris.
10. Any of the following within 14 days prior to initiation of study treatment:

    * Plasmapheresis;
    * Major surgery (kyphoplasty is not considered major surgery);
    * Radiation therapy;
    * Anti-myeloma drug therapy.
11. Received any investigational agents within 28 days or 5 half-lives (whichever is longer) prior to initiation of study treatment.
12. Conditions requiring chronic steroid or immunosuppressive treatment (eg, rheumatoid arthritis, multiple sclerosis, or lupus), which likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
13. Subjects may not receive corticosteroids (>10 mg/day of prednisone or equivalent) within 3 weeks prior to enrollment (use of steroidal inhalation aerosol for asthma is permitted).
14. Unable or unwilling to undergo antithrombotic prophylactic treatment.
15. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study, as determined by the Investigator.
16. Pregnant and/or breastfeeding females.
17. Known seropositive for or active viral infection with human immunodeficiency virus (HIV).
18. Known seropositive for or active viral infection with hepatitis B virus (HBV), with the following exceptions:

    * negative are eligible.
    * Subjects who had hepatitis B but have received an antiviral treatment and show non-detectable viral DNA for 6 months are eligible.
    * Subjects who are seropositive because of hepatitis B virus vaccine are eligible.
19. Known seropositive for or active viral infection with hepatitis C virus (HCV), with the following exception: Subjects who had hepatitis C but have received an antiviral treatment and show no detectable viral ribonucleic acid (RNA) for 6 months are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and/or recommended Phase 2 dose | Continuous up to one year

SECONDARY OUTCOMES:
Adverse events | Up to 5 years
Response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Reich, MD, Study Director — Triphase Research and Development I Corp
Locations (6):
- United States (4):
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chauhan D, Li G, Shringarpure R, Podar K, Ohtake Y, Hideshima T, Anderson KC. Blockade of Hsp27 overcomes Bortezomib/proteasome inhibitor PS-341 resistance in lymphoma cells. Cancer Res. 2003 Oct 1;63(19):6174-7. PMID 14559800
- [Background] Chauhan D, Singh AV, Ciccarelli B, Richardson PG, Palladino MA, Anderson KC. Combination of novel proteasome inhibitor NPI-0052 and lenalidomide trigger in vitro and in vivo synergistic cytotoxicity in multiple myeloma. Blood. 2010 Jan 28;115(4):834-45. doi: 10.1182/blood-2009-03-213009. Epub 2009 Nov 13. PMID 19965674
- [Background] Child JA, Morgan GJ, Davies FE, Owen RG, Bell SE, Hawkins K, Brown J, Drayson MT, Selby PJ; Medical Research Council Adult Leukaemia Working Party. High-dose chemotherapy with hematopoietic stem-cell rescue for multiple myeloma. N Engl J Med. 2003 May 8;348(19):1875-83. doi: 10.1056/NEJMoa022340. PMID 12736280
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Dexamethasone Prescribing Information. Roxane Laboratories Inc., Columbus, OH; Sep 2007. http://bidocs.boehringer-ingelheim.com/BIWebAccess/ViewServlet.ser?docBase= renetnt&folderPath=/Prescribing+Information/PIs/Roxane/Dexamethasone/Dexamethasone+Tablets+Solution+and+Intensol.pdf. Accessed 20 September 2013.
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Fermand JP, Katsahian S, Divine M, Leblond V, Dreyfus F, Macro M, Arnulf B, Royer B, Mariette X, Pertuiset E, Belanger C, Janvier M, Chevret S, Brouet JC, Ravaud P; Group Myelome-Autogreffe. High-dose therapy and autologous blood stem-cell transplantation compared with conventional treatment in myeloma patients aged 55 to 65 years: long-term results of a randomized control trial from the Group Myelome-Autogreffe. J Clin Oncol. 2005 Dec 20;23(36):9227-33. doi: 10.1200/JCO.2005.03.0551. Epub 2005 Nov 7. PMID 16275936
- [Background] Hideshima T, Chauhan D, Shima Y, Raje N, Davies FE, Tai YT, Treon SP, Lin B, Schlossman RL, Richardson P, Muller G, Stirling DI, Anderson KC. Thalidomide and its analogs overcome drug resistance of human multiple myeloma cells to conventional therapy. Blood. 2000 Nov 1;96(9):2943-50. PMID 11049970
- [Background] Howlader N, Noone AM, Krapcho M, et al. (eds). SEER Cancer Statistics Review, 1975 2009 (Vintage 2009 Populations), National Cancer Institute. Bethesda, MD, http://seer.cancer.gov/csr/1975_2009_pops09/. Accessed 20 September 2013.
- [Background] Kastritis E, Charidimou A, Varkaris A, Dimopoulos MA. Targeted therapies in multiple myeloma. Target Oncol. 2009 Jan;4(1):23-36. doi: 10.1007/s11523-008-0102-9. Epub 2009 Jan 17. PMID 19343299
- [Background] Kline JA, Wells PS. Methodology for a rapid protocol to rule out pulmonary embolism in the emergency department. Ann Emerg Med. 2003 Aug;42(2):266-75. doi: 10.1067/mem.2003.268. PMID 12883516
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Mitsiades N, Mitsiades CS, Poulaki V, Chauhan D, Richardson PG, Hideshima T, Munshi NC, Treon SP, Anderson KC. Apoptotic signaling induced by immunomodulatory thalidomide analogs in human multiple myeloma cells: therapeutic implications. Blood. 2002 Jun 15;99(12):4525-30. doi: 10.1182/blood.v99.12.4525. PMID 12036884
- [Background] Anderson KC, Alsina M, Bensinger W, Biermann JS, Chanan-Khan A, Cohen AD, Devine S, Djulbegovic B, Gasparetto C, Huff CA, Jagasia M, Medeiros BC, Meredith R, Raje N, Schriber J, Singhal S, Somlo G, Stockerl-Goldstein K, Tricot G, Vose JM, Weber D, Yahalom J, Yunus F; National Comprehensive Cancer Network. NCCN clinical practice guidelines in oncology: multiple myeloma. J Natl Compr Canc Netw. 2009 Oct;7(9):908-42. doi: 10.6004/jnccn.2009.0061. No abstract available. PMID 19878637
- [Background] Orlowski RZ, Nagler A, Sonneveld P, Blade J, Hajek R, Spencer A, San Miguel J, Robak T, Dmoszynska A, Horvath N, Spicka I, Sutherland HJ, Suvorov AN, Zhuang SH, Parekh T, Xiu L, Yuan Z, Rackoff W, Harousseau JL. Randomized phase III study of pegylated liposomal doxorubicin plus bortezomib compared with bortezomib alone in relapsed or refractory multiple myeloma: combination therapy improves time to progression. J Clin Oncol. 2007 Sep 1;25(25):3892-901. doi: 10.1200/JCO.2006.10.5460. Epub 2007 Aug 6. PMID 17679727
- [Background] Rajkumar SV, Harousseau JL, Durie B, Anderson KC, Dimopoulos M, Kyle R, Blade J, Richardson P, Orlowski R, Siegel D, Jagannath S, Facon T, Avet-Loiseau H, Lonial S, Palumbo A, Zonder J, Ludwig H, Vesole D, Sezer O, Munshi NC, San Miguel J; International Myeloma Workshop Consensus Panel 1. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1. Blood. 2011 May 5;117(18):4691-5. doi: 10.1182/blood-2010-10-299487. Epub 2011 Feb 3. PMID 21292775
- [Background] Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, San-Miguel JF, Blade J, Boccadoro M, Cavenagh J, Dalton WS, Boral AL, Esseltine DL, Porter JB, Schenkein D, Anderson KC; Assessment of Proteasome Inhibition for Extending Remissions (APEX) Investigators. Bortezomib or high-dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005 Jun 16;352(24):2487-98. doi: 10.1056/NEJMoa043445. PMID 15958804
- [Background] Richardson PG, Weller E, Jagannath S, Avigan DE, Alsina M, Schlossman RL, Mazumder A, Munshi NC, Ghobrial IM, Doss D, Warren DL, Lunde LE, McKenney M, Delaney C, Mitsiades CS, Hideshima T, Dalton W, Knight R, Esseltine DL, Anderson KC. Multicenter, phase I, dose-escalation trial of lenalidomide plus bortezomib for relapsed and relapsed/refractory multiple myeloma. J Clin Oncol. 2009 Dec 1;27(34):5713-9. doi: 10.1200/JCO.2009.22.2679. Epub 2009 Sep 28. PMID 19786667
- [Background] Richardson PG, Weller E, Lonial S, Jakubowiak AJ, Jagannath S, Raje NS, Avigan DE, Xie W, Ghobrial IM, Schlossman RL, Mazumder A, Munshi NC, Vesole DH, Joyce R, Kaufman JL, Doss D, Warren DL, Lunde LE, Kaster S, Delaney C, Hideshima T, Mitsiades CS, Knight R, Esseltine DL, Anderson KC. Lenalidomide, bortezomib, and dexamethasone combination therapy in patients with newly diagnosed multiple myeloma. Blood. 2010 Aug 5;116(5):679-86. doi: 10.1182/blood-2010-02-268862. Epub 2010 Apr 12. PMID 20385792
- [Background] Richardson PG, Jagannath S, Jakubowiak A, et al. Phase II Trial of Lenalidomide, Bortezomib, and Dexamethasone in Patients (pts) with Relapsed and Relapsed/Refractory Multiple Myeloma (MM): Updated Efficacy and Safety Data After > 2 Years of Follow-up. 2010b; ASH Annual Meeting Abstract #3049.
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Wells PS, Anderson DR, Rodger M, Ginsberg JS, Kearon C, Gent M, Turpie AG, Bormanis J, Weitz J, Chamberlain M, Bowie D, Barnes D, Hirsh J. Derivation of a simple clinical model to categorize patients probability of pulmonary embolism: increasing the models utility with the SimpliRED D-dimer. Thromb Haemost. 2000 Mar;83(3):416-20. PMID 10744147
- [Background] Wells PS, Anderson DR, Rodger M, Forgie M, Kearon C, Dreyer J, Kovacs G, Mitchell M, Lewandowski B, Kovacs MJ. Evaluation of D-dimer in the diagnosis of suspected deep-vein thrombosis. N Engl J Med. 2003 Sep 25;349(13):1227-35. doi: 10.1056/NEJMoa023153. PMID 14507948
- [Background] Velcade® (bortezomib) for Injection Prescribing Information. Millennium Pharmaceuticals Inc., Cambridge, MA; V-12-0388 02/13. http://www.velcade-hcp.com/previously-untreated-multiple-myeloma/dosing.aspx?gclid=CPD4lKn2tbsCFcU5Qgod9R0AdA.